CLINICAL TRIAL: NCT06289348
Title: Announcement of Rare Metabolic Diseases as Part of Systematic New-born Screening: the Experience of Phenylketonuria.
Brief Title: Announcement of Rare Metabolic Diseases in Systematic Newborn Screening: the Phenylketonuria Experience.
Acronym: ANNPHE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230240; 2023-A00970-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonuria
Keywords: presymptomatic announcement; systematic neonatal screening; rare diseases; genetic disease; phenylketonuria; care relationship; psychological trauma; psychological impact; parent-child bonding; parenthood
MeSH Terms: conditions — Phenylketonurias; Rare Diseases; Genetic Diseases, Inborn; Psychological Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- groupe 1: 60 parents of children screened for PKU. Each of them will be assessed using a socio-psychological questionnaire (7 days after the announcement) and the revised event impact scale (7 days, 4 and a half months).
  Interventions: Behavioral: socio-psychological questionnaire; Behavioral: revised event impact scale (IER-S)
- groupe 2: 25 parents from group 1. This smaller sample of 25 parents will be subjected to non-directive interviews (1 month after the announcement) and to the Stern interview (4 and a half months after the announcement).
  Interventions: Behavioral: socio-psychological questionnaire; Behavioral: revised event impact scale (IER-S); Other: Non directive interview; Other: Stern interview
- groupe 3: 15 doctors : interview
  Interventions: Other: semi-directive interview
- groupe 4: 5 midwifes : short interview
  Interventions: Other: semi-directive interview

INTERVENTIONS:
Behavioral: socio-psychological questionnaire — ton collecte socio-demographic variable
  Groups: groupe 1; groupe 2
Behavioral: revised event impact scale (IER-S) — 22 items assessed on a scale of frequency from 0 (not at all) to 4 (extremely)
  Groups: groupe 1; groupe 2
Other: Non directive interview — composed of a very broad opening sentence to encourage the parents' discourse
  Groups: groupe 2
Other: Stern interview — 54 questions to investigate the impact of the announcement and the parenthood construction
  Groups: groupe 2
Other: semi-directive interview — to propose ideas for improving and harmonizing practices
  Groups: groupe 3; groupe 4

SUMMARY:
The aims of this collaborative, interdisciplinary research project are to understand and describe the psychological impact of the announcement of a rare, serious disease present since birth and detected in the context of the systematic neonatal screening (DNS), in terms of the parents' experience, but also on the part of the medical team, in order to improve its process and the support it provides for the announcement of the diagnosis.

DETAILED DESCRIPTION:
In France, newborn screening for phenylketonuria (PKU) has been offered systematically, but not compulsorily, since 1970. This enables the disease to be treated at an early stage, with presymptomatic treatment. While treatment can significantly improve the prognosis of affected children, ensuring normal cognitive development without neurological sequelae, the announcement of the suspicion of the disease and confirmation of the diagnosis can be painful, even traumatic, for parents, due in particular to the very specific context of the DNS. The screening results are not available until 10 days after the baby's birth, and given the urgency of the treatment, the announcement is made by a telephone call to the families when they have already returned home with their asymptomatic newborn. This call was made by an unknown doctor from a center of reference or competence for rare diseases (in this case hereditary metabolic diseases, HMD), whom the parents did not know, and who asked them to come to his department as a matter of urgency. This disease is not visible at the time of diagnosis, although intoxication is already present. This research follows on from a pilot study2 which showed the traumatic nature of this call, which; for the families, means that in an instant they are thrust into the field of a rare, genetic and chronic disease; for the teams, means that the care relationship will continue until the end of the patient's adolescence. The aims of this collaborative, interdisciplinary research project are to understand and describe the psychological impact of the announcement of a rare, serious disease present since birth and detected in the context of the DNS, in terms of the parents' experience, but also on the part of the medical team, in order to improve its process and the support it provides for the announcement of the diagnosis.

The analysis will be carried out under the responsibility of the researcher, her thesis supervisor (Dr Marco Araneda, MCU / Université Paris-Cité) and her thesis co-supervisor (Pr Pascale de Lonlay, PU-PH / APHP and Université Paris-Cité).

1. Analysis of qualitative data :

   The interviews with the parents, doctors and midwives will be transcribed and then analysed using NVivo® software based on grounded theory methodology.
2. Analysis of quantitative data :

The data from the socio-psychological questionnaire will be analysed using simple, multidimensional descriptive statistics.

We will carry out an analysis of variance with repeated measures (IES-R) (time 1, time 2) to estimate the impact of time and care on the level of anxietý. A probabilitý level of 5% (p ≤ 0.05) will be considered́ significant for the results of the statistical tests. Statistical calculations will be performed using SPSS v.24 software, R y Mplus v. 8.3 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Parent or doctor of a child screened for PKU, born during the inclusion phase of the study
* Family's first exposure to PKU: the PKU child must be either the eldest or the first sibling to be diagnosed with PKU following neonatal screening

Exclusion Criteria:

* Failure to master the French language.
* Child screened is neither the eldest nor the first sibling to be screened.
* Refusal by the parents.
* Any other reason which, in the investigator's judgement, would impair the participants' ability to follow the study protocol, or the interpretation of interview data (e.g. the participating parent has a history of serious psychiatric pathology, one of the parents died at the child's birth, Couples in which one of the members suffers from a known decompensated psychiatric pathology at the time of recruitment. Couples where one of the members is under legal protection or a security measure, etc …).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parent(s) of children screened for PKU, doctors in charge of the announcement and midwives in charge of the NBS.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Psychological process linked to the announcement of inherited metabolic disease for the parents | 4 and a half months
  Identifying the psychological processes at work during and following the announcement of a child's illness (interview).
Psychological impact of the announcement of an inherited metabolic disease on the doctors' experience | 2 hours
  interview.
Measuring awareness of inherited metabolic diseases detected by midwives | 1 hour
  interview.

SECONDARY OUTCOMES:
Measure of the impact of the announcement on parents | 4 and a half months
  Psychometric scale (IER-S )

CONTACTS AND LOCATIONS:
Overall Officials: Céline BENSIMON, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No